CLINICAL TRIAL: NCT00510510
Title: A Randomized, Double-blind, Placebo Controlled, Parallel Group, Multi-center Study, to Assess the Safety and Tolerability of 28 Days Treatment With NVA237 (100 or 200 µg Once a Day) in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Safety and Tolerability of 28 Days Treatment With Glycopyrronium Bromide (NVA237) (100 or 200 µg Once a Day) in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CNVA237A2206
Record Dates: First submitted 2007-08-01; First posted 2007-08-02 (Estimated); Results first posted 2011-01-21 (Estimated); Last update posted 2012-05-21 (Estimated); Status verified 2012-05

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: COPD; glycopyrronium bromide; antimuscarinic
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Glycopyrrolate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (3):
- NVA237 100 µg (Experimental)
  Interventions: Drug: NVA237 100 µg
- NVA237 200 µg (Experimental)
  Interventions: Drug: NVA237 200 µg
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NVA237 100 µg — Dry powder inhalation once a day for up to 28 days
  Other Names: Glycopyrronium Bromide
  Arms: NVA237 100 µg
Drug: Placebo — Placebo to NVA237 dry powder inhalation once a day for up to 28 days
  Arms: Placebo
Drug: NVA237 200 µg — Dry powder inhalation once a day for up to 28 days
  Other Names: Glycopyrronium Bromide
  Arms: NVA237 200 µg

SUMMARY:
This study assessed the safety/tolerability of 28 days of treatment with NVA237 100 µg and 200 µg once a day, compared to placebo in patients with moderate or severe Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults aged 40 years or older
* Patients with moderate to severe COPD according to the GOLD Guidelines (2006)
* Patients who have smoking history of at least 10 pack years
* Patients with a post-bronchodilator Forced Expiratory Volume in One Second (FEV1) equal or greater than 30% of the predicted normal value and less than 80% of the predicted normal value, and post-bronchodilator FEV1/FVC less than 0.7 at visit 2
* Written informed consent by the patient prior to initiation of any study-related procedure

Exclusion Criteria:

* Patients requiring oxygen therapy on a daily basis for chronic hypoxemia, or who have been hospitalized for an exacerbation of their airways disease in the 6 weeks prior to visit 1 or during the screening period (up to visit 3).
* Patients who have had a respiratory tract infection within 6 weeks prior to visit 1 or during the screening period (up to visit 3).
* Patients with a history of asthma indicated by (but not limited to):

Blood eosinophil count > 400/mm3, onset of symptoms prior to age 40 years.

* Patients with a history of long QT syndrome or whose QTc measured at visit 1 is prolonged (more than 440 ms for males or more than 460 ms for females).
* Patients with a history of untoward reactions to sympathomimetic amines or inhaled medication or any component thereof.
* Patients who, in the judgment of the investigator have a clinically relevant laboratory abnormality or a clinically significant condition such as (but not limited to) unstable ischemic heart disease, left ventricular failure, long term prednisone therapy, history of myocardial infarction, arrhythmia, narrow-angle glaucoma, symptomatic prostatic hyperplasia, bladder-neck obstruction or moderate to severe renal impairment that might compromise patient safety or compliance, interfere with evaluation, or preclude completion of the study.
* History of malignancy of any organ system, treated or untreated, within the past 5 years whether or not there is evidence of local recurrence or metastases, with the exception of localized basal cell carcinoma of the skin.

Other protocol-defined inclusion/exclusion criteria may apply

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 281 (Actual)
Dates: Start 2007-08; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Chair — Novartis Pharmaceuticals
Locations (20):
- United States (15):
  - Novartis investigative site, Glendale, Arizona
  - Novartis investigative site, Phoenix, Arizona
  - Novartis investigative site, Wheat Ridge, Colorado
  - Novartis investigative site, Newark, Delaware
  - Novartis investigative site, Miami, Florida
  - Novartis investigative site, Tamarac, Florida
  - Novartis investigative site, River Forest, Illinois
  - Novartis investigative site, Overland Park, Kansas
  - Novartis investigative site, Saint Chares, Missouri
  - Novartis investigative site, Charlotte, North Carolina
  - Novartis investigative site, Portland, Oregon
  - Novartis investigative site, Spartanburg, South Carolina
  - Novartis investigative site, Union, South Carolina
  - Novartis investigative site, Fort Worth, Texas
  - Novartis investigative site, Houston, Texas
- Novartis investigative site, Rueil-Malmaison, France
- Novartis investigative site, Nuremberg, Germany
- Novartis investigative site, Arnhem, Netherlands
- Novartis investigative site, Barcelona, Spain
- Novartis investigative site, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Vogelmeier C, Verkindre C, Cheung D, Galdiz JB, Guclu SZ, Spangenthal S, Overend T, Henley M, Mizutani G, Zeldin RK. Safety and tolerability of NVA237, a once-daily long-acting muscarinic antagonist, in COPD patients. Pulm Pharmacol Ther. 2010 Oct;23(5):438-44. doi: 10.1016/j.pupt.2010.04.005. Epub 2010 Apr 21. PMID 20416390

RESULTS

PARTICIPANT FLOW:
Groups:
- NVA237 100 µg: NVA237 100 µg as a single dose dry powder inhaler (SDDPI), once a day in the morning for 28 days.
- NVA237 200 µg: NVA237 200 µg as a single dose dry powder inhaler (SDDPI), once a day in the morning for 28 days.
- Placebo: Matching placebo to NVA237 as a single dose dry powder inhaler (SDDPI), once a day in the morning for 28 days.
Period: Overall Study
Arm/Group | NVA237 100 µg | NVA237 200 µg | Placebo
Started | 92 | 98 | 91
Completed | 87 | 89 | 74
Not Completed | 5 | 9 | 17
Not completed — Adverse Event | 4 | 3 | 6
Not completed — Lack of Efficacy | 0 | 1 | 1
Not completed — Subjects no longer requires study drug | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 2 | 3
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 3 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NVA237 100 µg | NVA237 200 µg | Placebo | Total
Number analyzed (Participants) | 92 | 98 | 91 | 281
Age Continuous [Mean (Standard Deviation); unit: years] | 64.2 (7.93) | 62.6 (9.04) | 63.4 (9.44) | 63.4 (8.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 35 | 29 | 27 | 91
  Male | 57 | 69 | 64 | 190
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 17 | 15 | 11 | 43
  Not Hispanic or Latino | 72 | 79 | 76 | 227
  Unknown or Not Reported | 3 | 4 | 4 | 11
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 1
  Black or African American | 0 | 3 | 3 | 6
  White | 90 | 94 | 88 | 272
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 2 | 0 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Safety of Treatment With NVA237 in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease (COPD)
Description: The assessment of safety was based on adverse events, particularly those adverse events known to be associated to treatment with muscarinic antagonists. A summary of adverse events is presented with this outcome, additional details are provided in Adverse Events Sections.
Time Frame: 28 days
Measure: Number; unit: Participants
Arm/Group | NVA237 100 µg | NVA237 200 µg | Placebo
Number analyzed (Participants) | 92 | 98 | 91
Participants
  Total number of patients with any AE | 26 | 26 | 24
  Total number with any significant AE | 3 | 4 | 6

2. Secondary Outcome: Least Squares Means of Trough Forced Expiratory Volume in One Second (FEV1), by Day
Description: Forced expiratory volume maneuvers recorded using a calibrated spirometer. Trough forced expiratory volume in one second (FEV1) on Days 1 & 28 defined as the mean of the FEV1 values measured at 23 hours 15 minutes and 23 hours 45 minutes post-dose.
Time Frame: 28 Days
Measure: Least Squares Mean (Standard Error); unit: Liters
Arm/Group | NVA237 100 µg | NVA237 200 µg | Placebo
Number analyzed (Participants) | 92 | 98 | 91
Liters
  Trough FEV1 Day 1 | 1.465 (0.0152) | 1.480 (0.0149) | 1.334 (0.0154)
  Trough FEV1 Day 28 | 1.502 (0.0182) | 1.492 (0.0180) | 1.341 (0.0200)

ADVERSE EVENTS:
Arm/Group | NVA237 100 µg | NVA237 200 µg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/92 | 1/98 | 1/91
Other Adverse Events (participants affected / at risk) | 7/92 | 10/98 | 4/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 100 µg (N=92) | NVA237 200 µg (N=98) | Placebo (N=91)
Pneumonia (Infections and infestations) | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 — Chronic obstructive pulmonary disease exacerbation
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | NVA237 100 µg (N=92) | NVA237 200 µg (N=98) | Placebo (N=91)
Dry mouth (Gastrointestinal disorders) | 3 | 7 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 5 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.